CLINICAL TRIAL: NCT00296426
Title: Implementation and Evaluation of a Medical Reconciliation Protocol
Brief Title: Implementation and Evaluation of a Medical Reconciliation Protocol at Brigham and Women's Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Jeffrey Schnipper, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2005-P-002458/1
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Medication Reconciliation
Keywords: Adverse Drug Event; Inpatients; Outcome assessment
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

ARMS (2):
- Usual Care (No Intervention): control patients admitted to hospital floors received usual care
- Intervention (Experimental): computerized medication reconciliation tool and process redesign involving physicians, nurses, and pharmacists
  Interventions: Procedure: New technology - PAML

INTERVENTIONS:
Procedure: New technology - PAML
  Arms: Intervention

SUMMARY:
An incomplete understanding of patients' preadmission medications and failure to reconcile these with medications ordered in the hospital and at discharge are major, previously unappreciated, causes of adverse drug events (ADEs). The Joint Commission for Accreditation of Healthcare Organizations has now mandated a process for reconciling all medications at hospital admission and discharge. The best ways to implement medication reconciliation and the impact on patient outcomes are unknown. We, the researchers at at Brigham and Women's Hospital, will design and implement a medication reconciliation process with two major components: 1) information technology to integrate medication reconciliation into the current workflow at Brigham and Women's Hospital (BWH); and 2) process re-design involving physicians, nurses, and pharmacists to ensure that reconciliation takes place. We will then conduct a randomized controlled trial on the General Medical Service of BWH to evaluate the effects of this new process on reducing medication reconciliation errors with the potential to cause patient harm (potential ADEs).

DETAILED DESCRIPTION:
The primary outcome will be medication reconciliation errors with a potential for causing harm (potential ADEs). Secondary outcomes will include the different types of reconciliation errors, hospital length of stay, emergency department visits and hospital readmissions within 30 days of discharge, resident/nurse satisfaction, and compliance with the reconciliation process. To measure medication reconciliation errors, we will use a method similar to that suggested by the Massachusetts Coalition for the Prevention of Medical Errors. A study pharmacist, separate from the floor pharmacist, will determine each patient's preadmission medication regimen at the time of hospital discharge, using patient and family interviews and any additional information needed to validate the list. This list will then be compared with the preadmission medication list compiled by the intern to identify any errors in identifying preadmission medications. The list will also be compared with the admission and discharge medication orders in order to identify unexplained discrepancies. Questions will be resolved by communication between the study pharmacist and the ordering intern. Reports of all potential medication reconciliation errors will be presented in blinded fashion to two physician reviewers, who will judge whether a reconciliation error has taken place and its potential for harm. All medication reconciliation errors will be recorded, as well as each of the individual types: inaccuracies in the preadmission medication list, unexplained discrepancies with the admission medication orders, and unexplained discrepancies in the discharge orders. This methodology is similar to that used in other studies of medication errors conducted at BWH. This process will allow pharmacists to ethically report any problems to the medical team prior to discharge, while still allowing for a full measurement of medical errors. Hospital length of stay, emergency department visits, and hospital readmissions will be measured using hospital administrative data. Resident and nurse satisfaction and perceived quality of patient care will be measured using web-based surveys. Compliance with the reconciliation process will be measured by electronic tracking of the use and timing of: 1) PAML building and signing by the ordering intern, 2) reconciliation of all PAML medications within 24 hours of admission, and 3) reconciliation of the PAML and discharge medication orders by the ordering clinician at the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Must be inpatients on the General Medical Service at Brigham and Women's Hospital

Exclusion Criteria:

* Any other patients at BWH hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2006-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Schnipper JL, Hamann C, Ndumele CD, Liang CL, Carty MG, Karson AS, Bhan I, Coley CM, Poon E, Turchin A, Labonville SA, Diedrichsen EK, Lipsitz S, Broverman CA, McCarthy P, Gandhi TK. Effect of an electronic medication reconciliation application and process redesign on potential adverse drug events: a cluster-randomized trial. Arch Intern Med. 2009 Apr 27;169(8):771-80. doi: 10.1001/archinternmed.2009.51. PMID 19398689